CLINICAL TRIAL: NCT01104688
Title: Non Invasive in Vivo Evaluation of Abdominal Aorta Aneurysm Hemodynamics, Wall Stress, and Inflammation Using Magnetic Resonance Imaging
Brief Title: Non Invasive Imaging of Abdominal Aorta Aneurysm Hemodynamics and Wall Structure
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Nikolaj Eldrup, Counsultant MD PhD, Aarhus University Hospital
Other Study IDs: M-20100008
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: Abdominal Aortic Aneurysm; Wall Stress; Shear Stress; Inflammation; Magnetic Resonance Imaging
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Inflammation

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The development of the abdominal aorta aneurysm is multifactorial. Through use of magnetic resonance imaging without contrast, this study will look closely at flow, the stresses hereby induced, as well as signs of inflammation in the vessel wall.

DETAILED DESCRIPTION:
The etiology of the abdominal aorta aneurysm is complex and multi-factorial. Biomechanic and hemodynamic stress contributes to aneurysmal growth, and the relevance of inflammation is gaining in terms of pathological influence. The technical advances of imaging now enable one to utilize magnetic resonance in reconstructing aortal blood flow. Newer post-imaging software then enables one to perform complex data analysis, wherein shear and wall-stress can be calculated. The goal of this study is to analyze the aneurysms of twenty patients. Values will be obtained for shear and wall stress. Additionally, the utilization of short tau wave inversion recovery (STIR) sequences will be performed to evaluate the presence or absence of acute edema and inflammation of the region. It should also be noted that particular attention will be placed on the so-called "neck" of the aneurysm, where the aneurysm typically tapers into what is often regarded as normal aortic tissue. This region is important for both the placement of a surgical bypass prosthesis or a deployed stent graft.

ELIGIBILITY:
Inclusion Criteria:

* Infrarenal abdominal aorta aneurysm (AAA)

Exclusion Criteria:

* Lack of signed, informed consent
* Pacemaker or other implanted metal prostheses
* Claustrophobia
* Dementia
* Diabetes Mellitus
* Thoracoabdominal aorta aneurysm, per Crawford/Safi criteria
* Ehlers-Danlos, Marfans, or other diagnosed connective tissue disease

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty patients diagnosed with an infrarenal abdominal aorta aneurysm will be selected from our clinical database.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Left ventricular longitudinal strain for perioperative cardiac monitoring in aortic aneurysm surgery using transthoracic 2-dimensional echocardiography: a a feasibility and repeatability study.feasibility and repeatability study. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jacob W Budtz-Lilly, MD, Principal Investigator — Aarhus University Hospital Skejby, Department of cardiothoracic and vascular surgery
Locations (1):
- Aarhus University, Skejby Hospital, Department of cardiothoracic and vascular surgery & MR-center, Aarhus, Denmark